CLINICAL TRIAL: NCT07025954
Title: Planned Delivery at 37 Versus 36 Weeks in Pregnancies Complicated byPlacenta Previa and Accreta: A Randomized Controlled Trial
Brief Title: Planned Delivery at 37 Versus 36 Weeks in Pregnancies With Placenta Previaand Accreta
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, wangzhijian, Professor, MD, PhD, The Third Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB(2025)-061
Record Dates: First submitted 2025-05-21; First posted 2025-06-18 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Placenta Previa; Placenta Accreta Spectrum; Antepartum Bleeding; Emergency Cesarean Section; Preterm Birth Complication
MeSH Terms: conditions — Placenta Previa; Placenta Accreta | interventions — Cesarean Section

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 37-week group (Experimental): Subjects were randomized 1:1 at 28-34 weeks. 37-week group: planned delivery at 37 0/7-37 6/7 weeksof gestation.
  Interventions: Procedure: Cesarean delivery
- 36-week group (Active Comparator): Subjects were randomized 1:1 at 28-34 weeks. 36-week group: planned delivery at 36 0/7-36 6/7 weeksof gestation.
  Interventions: Procedure: Cesarean delivery

INTERVENTIONS:
Procedure: Cesarean delivery — All patients were delivered via cesarean section with standardized perioperative management, including preoperative preparation (e.g., autologous bloodreserve, corticosteroid administration for foetal lungmaturation, etc.), surgical approach, and postoperative care.
  Conservative management (intentional placental retention in situ with local resection and pelvic devascularization) was primarily employed, while peripartum hysterectomy was reserved for those with extensive invasion or failed conservative treatment.

SUMMARY:
Current clinical practice guidelines recommend planned cesarean delivery(CD) at 34-37 weeks of gestation in pregnant women with placenta previa and accreta. Preterm birth may lead to neonatal immaturity, while laterCD may increase the risk of severe hemorrhage and surgery complications. Retrospective studies have shown that indicated CD occurs in approximately1/3 of patients before 36 weeks, with the main trigger being antepartum hemorrhage. However, the risk of antepartum hemorrhage is lower after 36 weeks. Recent study showed that delivery shifted from 34-36 weeks to 37 weeks did not increase therisk of maternal intraoperative/postoperative hemorrhage and emergency CD. To further validate this, we propose to conduct a randomized controlled study comparing the effect of planned delivery management strategies at 37 0/7-37 6/7 weeks of gestation with those at 36 0/7-36 6/7 weekson maternal and fetal outcomes. The aim of this study is to explore whether planned delivery up to 37 weeks in pregnant women with placenta previa and accreta improves neonatal outcomes without increasing maternal obstetric risks.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label, randomized controlled trial, which aims to determine the optimal delivery timing for pregnant women with placenta previa and accreta. Participants were stratified by centers and randomly assigned in 1:1 at 28-34 weeks of gestation. Opaque sealed envelopes used to mask randomization sequences. The primary efficacy outcome is the composite neonatal morbidity rate, while the primary safety outcome is intraoperative estimated blood loss (EBL) during cesarean delivery. Secondary outcomes include the incidence of unplanned cesarean delivery, hysterectomy rate, maternal ICU admission, total packed red blood cell transfusion (units), operative duration (hours), surgical complications, unplanned reoperation rate, postpartum morbidity, and neonatal NICU admission. Statistical analyses will be performed based on the intent-to-treat (ITT) principle using the full analysis set (FAS), with a supportive per-protocol (PP) analysis. The statisticians will remain blinded to group assignments through coded data until the final analysis is completed.

ELIGIBILITY:
Inclusion Criteria:

* 28-34 weeks of gestation.
* Both ultrasound and MRI indicate placenta previa with placenta accreta spectrum (PAS).
* Planned to undergo cesarean delivery at the participating study hospitals.
* Agree to participate and sign the informed consent form.

Exclusion Criteria:

* Multiple gestation.
* Other obstetric complications (e.g., preeclampsia, vasa previa), and severe maternal medical conditions (e.g., uncontrolled diabetes, progressive cardiovascular disease, active systemic lupus erythematosus, liver cirrhosis).
* Major uterine structural anomalies (e.g., uterine didelphys, Uterine tumors ≥5 cm).
* Estimated fetal weight <3rd percentile for gestational age, major congenital anomalies, intrauterine fetal demise.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Composite neonatal morbidity | Within 30 days after childbirth
  The Composite neonatal morbidity was defined as any of the following: admission to the Neonatal Intensive Care Unit (NICU), need for mechanical ventilation (MV), Respiratory Distress Syndrome (RDS), Transient Tachypnea of Newborn (TTN), Necrotizing Enterocolitis (Necrotizing Enterocolitis), and necrotizing Enterocolitis (NEC). Syndrome (RDS), Transient Tachypnea of Newborn (TTN), Necrotizing Enterocolitis (NEC), Intraventricular Hemorrhage (IVH), Septicemia (S), and Necrotizing Enterocolitis (NE). IVH), sepsis (Sepsis), and neonatal death. Evaluator blinding was used to ensure the objectivity of the assessment, and the pediatrician responsible for assessing neonatal complications was unaware of the grouping information.
Intraoperative Estimated Blood Loss (EBL) | From surgery initiation to 24 hours postoperatively
  Intraoperative EBL was calculated during delivery using a combined gravimetric and volumetric method: all surgical gauzes and drapes were weighed before the procedure (preoperative weight), and blood-soaked gauzes and drapes were weighed postoperatively (postoperative weight); the baseline fluid volume in the suction canister was recorded before amniotic fluid aspiration, and the total volume was recorded immediately after completion of amniotic fluid aspiration (amniotic fluid volume = post-aspiration volume - baseline volume). The final EBL （ml）was calculated as: (postoperative weight - preoperative weight) + (total suctioned volume - amniotic fluid volume - irrigation fluid volume).

SECONDARY OUTCOMES:
Incidence of unplanned cesarean delivery | Immediately after procedure
  Unplanned cesarean delivery refers to all cesarean sections performed prior to the gestational age specified in the study protocol, including indications such as uncontrolled antepartum hemorrhage, preterm labor, fetal distress, and other complications requiring delivery before the designated gestational age.
Rate of Hysterectomy | Within 30 days after childbirth
  Hysterectomy refers to total or subtotal hysterectomy performed due to refractory hemorrhage during cesarean delivery or postpartum conservative treatment, excluding hysterectomies performed for conditions such as uterine tumors.
Perioperative RBC transfusion (U) | Perioperatively
  The cumulative unit of packed RBC transfused during hospitalization for delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Wang, MD, PhD, Principal Investigator — The Third Affiliated Hospital of Guangzhou Medical University
Locations (6):
- China (6):
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - West China Second University Hospital, Sichuan University, Chengdu, Sichuan
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangzhou Women and Children's Medical Center, Guangzhou

IPD SHARING:
Plan to Share IPD: No